CLINICAL TRIAL: NCT01957553
Title: Investigating the Safety and Performance of a New 2-piece Ostomy Product Compared With SenSura Click in 130 Subjects With an Ileostomy.
Brief Title: Investigating the Safety and Performance of a New 2-piece Ostomy Product Compared With SenSura Click 2-piece
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP243
Record Dates: First submitted 2013-10-01; First posted 2013-10-08 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence 1, First Coloplast Test product (Experimental): Subjects first allocated to Coloplast Test product will after cross-over test SenSura
  Interventions: Device: Coloplast test product; Device: SenSura
- Treatment seqence 2; First SenSura (Experimental): Subjects first allocated to SenSura will after cross-over test Coloplast Test product
  Interventions: Device: Coloplast test product; Device: SenSura

INTERVENTIONS:
Device: Coloplast test product — Coloplast test product is a newly developed 2-piece ostomy appliance
Device: SenSura — SenSura is the commercial available CE-marked SenSura Click 2-piece ostomy appliance from Coloplast A/S
  Other Names: SenSura Click; SenSura Standard 2-piece

SUMMARY:
The aim of the current investigation is to investigate the performance of a new 2-piece ostomy product

DETAILED DESCRIPTION:
The present investigation aims at testing the performance and safety of a new 2-piece ostomy product.

ELIGIBILITY:
Inclusion Criteria:

* 1.Have given written informed consent and letter of authority (DK only)
* 2.Be at least 18 years of age and have full legal capacity.
* 3.Be able to handle the products her/himself
* 4.Have an ileostomy with a diameter between 10 and 40 mm.
* 5.Have had their ostomy for at least three months.
* 6.Be willing to use minimum 2 base plates every week
* 7.Currently use 2-piece flat mechanical coupling product with open bag 8
* 11.Negative result of a pregnancy test for women of childbearing age (only DK)

Exclusion Criteria:

* 1.Currently receiving or have within the past 2 months received radio- and/or chemotherapy.
* 2.Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
* 3.Is pregnant or breastfeeding.
* 4.Is participating in other interventional clinical investigations or have previously participated in this investigation
* 5.Has participated in the previous explorative study CP234
* 6.
* 7.Known hypersensitivity towards any of the test products
* 8.Currently suffering from peristomal skin problems (i.e.bleeding or red and broken skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Coloplast A/S
Locations (17):
- Imelda Hospital Bonheiden, Bonheiden, Belgium
- Denmark (6):
  - Aabenraa Stomi Ambulatorie, Sygehus Sønderjylland, Aabenraa
  - Coloplast A/S, Humlebæk
  - Stomiambulatoriet, Kolding Sygehus, Kolding
  - Stomiambulatoriet A5, Odense Hospital, Odense C
  - Kirurgisk ambulatorium/Stomiambulatoriet OUH, Svendborg
  - Vejle Sygehus, Stomiambulatoriet B120, Vejle
- QPS Netherlands, Groningen, Netherlands
- Norway (2):
  - Gastrokirurgisk Sekjon, Kirurgisk Klinikk Haugesund Sjukhus, Haugesund
  - Helse Nordbyen, Larvik
- Sweden (7):
  - Länssjukhhuset gävle, Stomimottagningen, Gävle
  - Kirug kliniken Centralsjukhuset, Karlstad
  - Kirurgens Mottagning, Malmo
  - Capio St. Görans Sjukhus AB, kirurgkliniken, Stockholm
  - Södersjukhuset, Stockholm
  - karolinska Universitetssjukhuset Solna Stomimottagningen, Stockholm
  - Stomimottagningen Centrllasarette i Västerås, Västerås

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited from Coloplast user data base, from hospital sites and stoma care sites.
Pre-assignment Details: 130 subjects were randomised, however 3 of these were not exposed to a product and where not included in the safety population. The participant flow below is generated based on the safety population.
Groups:
- Treatment Sequence 1, First Coloplast Test Product, the SenSur: Subjects first allocated to Coloplast Test product will after cross-over test SenSura
  Coloplast test product: Coloplast test product is a newly developed 2-piece ostomy appliance
  SenSura: SenSura is the commercial available CE-marked SenSura Click 2-piece ostomy appliance from Coloplast A/S
- Treatment Seqence 2; First SenSura the Coloplast Test Product: Subjects first allocated to SenSura will after cross-over test Coloplast Test product
  Coloplast test product: Coloplast test product is a newly developed 2-piece ostomy appliance
  SenSura: SenSura is the commercial available CE-marked SenSura Click 2-piece ostomy appliance from Coloplast A/S
Period: Test Period 1 (21 +- 1 Days)
Arm/Group | Treatment Sequence 1, First Coloplast Test Product, the SenSur | Treatment Seqence 2; First SenSura the Coloplast Test Product
Started | 61 | 66
Completed | 54 | 63
Not Completed | 7 | 3
Not completed — Lack of Efficacy | 2 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — screen failure | 1 | 0
Period: Test Period 2 (21 +- 1 Days)
Arm/Group | Treatment Sequence 1, First Coloplast Test Product, the SenSur | Treatment Seqence 2; First SenSura the Coloplast Test Product
Started | 54 | 63
Completed | 51 | 56
Not Completed | 3 | 7
Not completed — Adverse Event | 1 | 3
Not completed — Lack of Efficacy | 1 | 2
Not completed — completed early by mistake | 0 | 1
Not completed — device deficiency without AE | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are summarized with the subjects included in the ITT population. Two subjects where exposed to a product but did not register any endpoint data. These subjects are only found in the safety population.
Groups:
- All Subjects: baseline data are summarized for all subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Preference
Description: The subjects were asked which product they preferred (the Test product or SenSura) at the end of the investigation. The preference result shows the percentage of subjects preferring either the Test product or SenSura.
Time Frame: 21+1 days
Population: The ITT population was constituted by all randomized subjects with valid informed consent who had applied at least one test product and had valid information for the primary endpoint preference, or valid information for at least one product with respect to one of the secondary endpoints., who included all subject who contributed with endpoint data
Measure: Number; unit: percentage of participants
Arm/Group | Coloplast Test Product | SenSura
Number analyzed (Participants) | 114 | 114
percentage of participants | 65 | 35

ADVERSE EVENTS:
Time Frame: 42+/- 3 days
Groups:
- Test Product: Safety data for subjects exposed to the test product
- SenSura: Safety data for subjects exposed to SenSura
Arm/Group | Test Product | SenSura
Serious Adverse Events (participants affected / at risk) | 4/124 | 1/120
Other Adverse Events (participants affected / at risk) | 27/124 | 22/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=124) | SenSura (N=120)
pain in chest (Cardiac disorders) | 1 (1) | 0 (0) — not related to device
rectal bleeding/inflammtion of the intestine (Gastrointestinal disorders) | 1 (1) | 0 (0) — unlikely related to device
Sclerosing angiomatoid nodlar tranformation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Not related to device
A cystic lesion in operation area (Surgical and medical procedures) | 1 (1) | 0 (0) — Not related to device
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Not related to device
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Not related to device
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=124) | SenSura (N=120)
peristomal skin irritation (Skin and subcutaneous tissue disorders) | 27 (46) | 22 (35) — The adverse events are related to the device. Related adverse events includes the adverse events in the categories 'unlikely related', possibly related', 'probably related' and 'definitely related'.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less